CLINICAL TRIAL: NCT04801771
Title: Effects of Hypoglossal Nerve Stimulation on Cognition and Language in Down Syndrome and Obstructive Sleep Apnea
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Inspire Medical Systems, Inc. (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-003; 1U01DC019279-01 (NIH)
Record Dates: First submitted 2020-12-15; First posted 2021-03-17 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Down Syndrome; Obstructive Sleep Apnea
Keywords: Hypoglossal nerve stimulation
MeSH Terms: conditions — Down Syndrome; Sleep Apnea, Obstructive | interventions — Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: Hypoglossal Nerve Stimulation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Subjects implanted with Inspire UAS System (Experimental): Subjects who meet eligibility criteria will be implanted with the Inspire Upper Airway Stimulation (UAS) System.
  Interventions: Device: Inspire Upper Airway Stimulation (UAS) System

INTERVENTIONS:
Device: Inspire Upper Airway Stimulation (UAS) System — The Inspire UAS System is an implantable device that provides hypoglossal nerve stimulation for the treatment of obstructive sleep apnea.
  Other Names: Hypoglossal nerve stimulation

SUMMARY:
This study is a prospective, single-arm study conducted under a common implant and follow-up protocol. The objective will be to follow fifty-seven (57) adolescents and young adults (10-21 years of age), with Down syndrome, moderate to severe sleep apnea, and post-adenotonsillectomy, for 12 months after undergoing implant of the Inspire Upper Airway Stimulation (UAS) System. The study is being conducted in order to evaluate objective change in cognition and expressive language after implant and therapy with the Inspire UAS System.

DETAILED DESCRIPTION:
This study is a prospective, single-arm study conducted under a common implant and follow-up protocol. The objective will be to follow fifty-seven (57) adolescents and young adults (10-21 years of age), with Down syndrome, moderate to severe sleep apnea, and post-adenotonsillectomy, for 12 months after undergoing implant of the Inspire Upper Airway Stimulation (UAS) System. The study is being conducted in order to evaluate objective change in cognition and expressive language after implant and therapy with the Inspire UAS System.

Prior to implant subjects will be required to meet eligibility criteria, complete quality of life questionnaires and undergo neurocognitive testing (NCT) and expressive language sampling. Eligibility criteria will be determined via review of medical records, an in-lab polysomnography (sleep study), and a drug-induced sleep endoscopy (DISE).

After implant of the Inspire UAS System, subjects will undergo five (5) study visits. Four (4) of the visits will include an in-lab sleep study (PSG). Follow-up expressive language sampling and neurocognitive testing will be performed at 6 months post-implant. Follow-up quality of life questionnaires will be completed at 12 months post-implant.

Subjects will conclude their participation in the study at the end of their 12 month study visit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Down syndrome
* Age 10-21 years
* Prior adenotonsillectomy
* Severe OSA (AHI > 10, AHI < 50, no more than 25% AHI attributable to central events) based on prior in-lab PSG performed after adenotonsillectomy and within 18 months of enrollment
* Approval from at least two of the three physician reviewers based upon the results of a routine drug-induced sleep endoscopy (DISE) having occurred within 12 months of enrollment
* Subjects must have either tracheotomy or be ineffectively treated with CPAP due to non-compliance, discomfort, un-desirable side effects, persistent symptoms despite compliance use, or refusal to use the device
* Children and their parents/guardians must be willing to have stimulation hardware permanently implanted, and be willing to participate in follow-up visits, postoperative PSG, and questionnaire completion
* Children's parents/guardians must complete a questionnaire confirming that their child is capable of communicating feelings of pain or discomfort. They must also confirm they are able to assess their child for adverse effects related to device implantation
* Children and their parents/guardians must be proficient in English

Exclusion Criteria:

* Body mass index (BMI) above the 95th percentile for subject's age
* Circumferential airway collapse at the level of the velopharynx observed during DISE
* Other medical conditions resulting in medical instability (eg. congestive heart failure, recent open heart surgery, immunosuppression, or chronic lung disease or aspiration)
* Presence of another medical condition requiring future magnetic resonance imaging (MRI) of the chest
* Patients with another implantable device which could interact unintentionally with the Inspire system
* Any contraindication for general anesthesia
* History of bleeding or clotting disorders and those on blood thinning or NSAID medications for the week prior to implantation surgery. Subjects will be asked to refrain from the use of NSAIDS for two weeks after implantation or any revision surgeries
* Subject is currently taking muscle relaxant medication
* Life expectancy less than 12 months
* Subject's inability to communicate pain or discomfort to their caretaker/parent, based on parental or investigator assessment
* Nonverbal candidates will be excluded due to an inability to complete testing procedures including expressive language sampling
* Subjects with a co-occurring diagnosis of autism spectrum disorder
* Subjects that have a positive β-HCG
* Subjects deemed unfit for participation by the investigator for any other reason

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 57 (Estimated)
Dates: Start 2021-06-24 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in intelligence using the Kaufman Brief Intelligence Scale (KBIT-2) | 6 Months post-implant
  Change in the Intelligence Quotient Standard Score of at least 0.5 standard deviation from baseline
Change in attention using the Wechsler Intelligence Scale | 6 Months post-implant
  Change in Cancellation scaled score of at least 0.5 standard deviation from baseline
Change in processing speed using the Cambridge Neuropsychological Test Automated Battery (CANTAB) | 6 Months post-implant
  Change in RTIFMDRT and RTIFMDMT raw scores of at least 0.5 standard deviation from baseline
Change in executive functioning using the Delis-Kaplan Executive Functioning System (DKEFS) | 6 Months post-implant
  Change in Category Functioning scaled score of at least 0.5 standard deviation from baseline
Change in learning and memory using the Cambridge Neuropsychological Test Automated Battery - Paired Associates Learning | 6 Months post-implant
  Change in PAL-TEA raw score of at least 0.5 standard deviation from baseline
Change in language using Expressive Language Sampling | 6 Months post-implant
  Change in % of unintelligible C-units, number of different word roots and mean length of C-units in morphemes of at least 0.5 standard deviation from baseline

SECONDARY OUTCOMES:
Rate of procedure and device-related adverse events | Implant through 12 Months post-implant
  Procedure and device-related adverse events will be collected in order to profile the safety of hypoglossal nerve stimulation in adolescents. Number and percent of procedure and device-related adverse events will be reported
Change in Obstructive Sleep Apnea (OSA) | 3, 6, 12 Months post-implant
  Change in sleep apnea will be measured using standard in-lab PSG measures including oxygen level, partial and complete airway obstruction, and arousals. Improvement will be defined as a 50% or more decrease in AHI.
Change in quality of life as measured by OSA-18 and ESS-CHAD questionnaires | 12 months post-implant
  Quality of life improvements will be measured using the OSA-18 and ESS-CHAD. Mean scores for each questionnaire will be reported at baseline and 12 months post-implant.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Hartnick, MD, Principal Investigator — The Massachusetts Eye and Ear Infirmary
Locations (8):
- United States (8):
  - Children's Healthcare of Atlanta/ Emory University School of Medicine, Atlanta, Georgia
  - Massachusetts General Hospital (Mass Eye & Ear Infirmary), Boston, Massachusetts
  - Cincinnati Childrens Hospital, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas Southwestern/Children's Hospital of Dallas, Dallas, Texas
  - Children's Hospital of the King's Daughters/East Virginia Medical School, Norfolk, Virginia
  - University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No